CLINICAL TRIAL: NCT06570070
Title: Effectiveness of Artificial Intelligence (AI)-Powered Chatbot vs. Human Counselors in Smoking Cessation
Brief Title: AI-powered Chatbot vs. Human Counselors in Smoking Cessation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AI-powered cessation support
Record Dates: First submitted 2024-08-16; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Smoking Cessation; Mobile Health
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AI support group (Experimental): AI-powered chatbot support+ 5A's/5R's advice + health warning leaflet+ Self-help booklet
  Interventions: Behavioral: 5A's/5R's advice; Other: Brief leaflet on health warning and smoking cessation; Other: Self-help smoking cessation booklet; Behavioral: AI-powered chatbot support
- Counselor support group (Experimental): Counselor individual support+ 5A's/5R's advice + health warning leaflet+ Self-help booklet
  Interventions: Behavioral: 5A's/5R's advice; Other: Brief leaflet on health warning and smoking cessation; Other: Self-help smoking cessation booklet; Behavioral: Counselor individual support
- Control group (Active Comparator): 5A's/5R's advice + health warning leaflet+ Self-help booklet
  Interventions: Behavioral: 5A's/5R's advice; Other: Brief leaflet on health warning and smoking cessation; Other: Self-help smoking cessation booklet

INTERVENTIONS:
Behavioral: 5A's/5R's advice — 5A's (Ask, Advise, Assess, Assist, Arrange) for smokers who are ready to quit, and 5R's (relevance, risks, rewards, roadblocks, and repetition) for smokers who are not ready to quit.
Other: Brief leaflet on health warning and smoking cessation — The contents of the leaflet include the absolute risk of smoking, diseases caused by active and second-hand smoking, horrible pictorial warnings of the health consequences of active and second-hand smoking, and the benefits of quitting.
Other: Self-help smoking cessation booklet — The contents include information about the benefits of quitting, methods to quit, how to handle withdrawal symptoms, misperceptions of quitting, etc.
Behavioral: AI-powered chatbot support — Participants will receive three months of AI-powered chatbot, equipped with personalized interactions and real-time support, via WeChat.
  Arms: AI support group
Behavioral: Counselor individual support — Participants will receive three months of counselor-led individual support via WeChat. The regular messages and instant messaging on psychosocial support aim to provide cessation advice, increase self-efficacy and confidence, and social support and behavioral capacity of quitting.
  Arms: Counselor support group

SUMMARY:
This study aims to explore the feasibility and preliminary effectiveness of AI-powered chatbot support in community smokers.

DETAILED DESCRIPTION:
Smoking cessation remains one of the most significant public health challenges worldwide, with tobacco use being a leading cause of preventable death and disease. Despite extensive efforts, the success rates of smoking cessation programs remain low, necessitating innovative approaches to support individuals in their journey to quit smoking. Recently, artificial intelligence (AI) has opened new possibilities in healthcare, including the development of AI-powered chatbots that assist individuals in behavior change, such as quitting smoking.

This randomized controlled trial aims to investigate the effectiveness of AI-powered chatbot that simulates human counselors, compared to traditional human counseling in promoting smoking cessation among community smokers. The AI-powered chatbot, equipped with personalized interactions and real-time support, offers scalable and cost-effective assistance, potentially making it an accessible alternative to human counseling. However, human counselors provide empathy, tailored advice, and a nuanced understanding of human behavior that AI may not fully replicate. This study will explore which approach is more effective in helping individuals achieve long-term smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 and above, reside in Zhuhai for the next 6 months;
2. smoke at least 1 cigarette or use e-cigarettes daily;
3. Having a smartphone and a WeChat account, being able to use WeChat skillfully.

Exclusion Criteria:

1. Smokers who have communication barrier (either physically or cognitively);
2. Smokers who are currently participating in other SC programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical validated quit rate at 6 months follow-up | 6 months follow-up
  The primary outcomes are biochemically validated quit rate (exhaled carbon monoxide < 4 ppm or salivary cotinine < 30 ng/ml)

SECONDARY OUTCOMES:
Biochemical validated quit rate at 3 months follow-up | 3 months follow-up
  biochemically validated quit rate (exhaled carbon monoxide < 4 ppm or salivary cotinine < 30 ng/ml)
Self-reported 7-day point prevalence quit rate | 3 and 6 months follow-up
  Self-reported 7-day point prevalence quit rate in the two groups
Smoking reduction rate | 3 and 6 months follow-up
  Rate of smoking reduction by at least half of baseline amount in the two groups
Eligibility rate | baseline
  the percentage of eligible smokers out of the total number of smokers screened
Consent rate | baseline
  the percentage of eligible smokers who agree to participate out of the total number of eligible smokers
Percentage of Participant Engagement with E-Messages and Counselor Chats | 3 months follow-up
  This outcome measures the percentage of participants who engage with the intervention by reading e-messages and responding to counselor chat messages at least once during the 3-month follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Normal University, Zhuhai, Guangdong, China